CLINICAL TRIAL: NCT05648123
Title: Effectiveness of Supportive Psychotherapy Through Internet-Based Teleconsultation on Psychological and Somatic Symptoms, Neutrophil-Lymphocyte Ratio, and Heart Rate Variability in Post Covid-19 Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Dika Iyona Sinulingga, SpPD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22111301
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Psychotherapy (Experimental): supportive psychotherapy will be given in the form of an online group for 3 times a week with a duration of psychotherapy ranging from 1 - 2 hours per session
  Interventions: Behavioral: Supportive Psychotherapy
- Education (Active Comparator): education about post covid-19 syndrome will be given in the form of an online group for 3 times a week with a duration about 1 - 2 hours per session
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Supportive Psychotherapy — Supportive psychotherapy is a treatment that uses direct measures to ameliorate symptoms and to maintain, restore or improve self-esteem, ego function, and adaptive skills

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of supportive psychotherapy in post covid-19 syndrome patients. The main questions it aims to answer are:

1. What is the effect of supportive psychotherapy on psychological and somatic symptoms in post covid-19 syndrome patients?
2. What is the effect of supportive psychotherapy on the neutrophil lymphocyte ratio in post covid-19 syndrome patients?
3. What is the effect of supportive psychotherapy on heart rate variability in post covid-19 syndrome patients?

Participants will be given supportive psychotherapy in the form of an online group for 3 times a week with a duration of psychotherapy ranging from 1 - 2 hours per session.

Researchers will compare the supportive psychotherapy group to education group as control. The control group will be given education about Post Covid-19 syndrome in the form of an online group for 3 times a week with a duration of around 1 - 2 hours per session.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Patients confirmed positive for SARS CoV-2 by molecular testing (SARS CoV-2 RT-PCR, naso-oropharyngeal swab) at least 3 months before recruitment, with symptoms and effects lasting for at least 2 months and not explained by alternative diagnoses other
* Patients with or without comorbidities: diabetes mellitus, hypertension, tuberculosis, asthma, chronic obstructive pulmonary disease, chronic kidney disease, heart disease, chronic liver disease, malignancy, nervous system disease, patients with vulnerability, patients with disabilities.
* Patients can communicate and are willing to be interviewed, fill out questionnaires and psychotherapy.
* The patient is willing to fill out and sign an informed 1 sheet of consent to participate in the study

Exclusion Criteria:

* Psychosis
* Can not access internet for psychotherapy
* Not willing to take part in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Pyschological and somatic symptoms | Change from baseline SCL-90 questionnaire at 1 week
  Measured with SCL-90 questionnaire. Minimum score is 0, maximum score is 360. Higher scores mean worse outcome
Neutrophil Lymphocyte Ratio (NLR) | Change from baseline NLR at 1 week
  Measured by calculating the value of the ratio of neutrophils and lymphocytes based on blood sampling
Heart Rate Variability | Change from baseline SDNN at 1 week
  Measured by assessing SDNN by using Photoplethysmograph SA-3000P

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia